CLINICAL TRIAL: NCT04738773
Title: Double Blind 12-week Controlled Experiment With Two Groups of Pathological Gamblers, One Taking Active Drug (Naltrexone) and the Other Receiving Placebo.Patters Patterns of Visual Tracking Will be Acessed on Both Groups Prior and During Tratment in Order to Predict Treatment Response
Brief Title: RCT for Gambling and Naltrexone, Using Use Eye-tracking Analysis to Predict Treatment Response
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Hermano Tavares, Associate Profssor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gambling Natrexone ET
Record Dates: First submitted 2021-01-31; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Eye Tracking; Gambling Disorder; Naltrexone
MeSH Terms: conditions — Gambling | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients receiving Naltrexone (Active Comparator)
  Interventions: Drug: Naltrexone
- Patients receiving Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — On the active drug group, naltrexone will be prescribed on flexible dose mode, receiving 50mg per day on the first week, with an increase of 25mg each week until a maximum of 200 mg per day or as much as tolerated by the patient.
  Arms: Patients receiving Naltrexone
Drug: Placebo — Placebo
  Arms: Patients receiving Placebo

SUMMARY:
The primary objective of this study is to determine whether favorable response to naltrexone orally taken in treatment of GD can be predicted by patterns of visual scanning, assessed by eye-tracking technology before, at the start and throughout gambling treatment with naltrexone.

DETAILED DESCRIPTION:
The study will be a double blind 12-week controlled trial with two groups, one taking active drug (naltrexone) and the other receiving placebo. Patients on both groups will be assessed for GD symptoms and severity, major comorbid psychiatric disorders and related psychopathology (impulsivity, craving and locus of control), and eye-tracking patterns prior to and one hour after the administration of the first dose, one week after and at treatment completion.

On the active drug group, naltrexone will be prescribed on flexible dose mode, receiving 50mg per day on the first week, with an increase of 25mg each week until a maximum of 200 mg per day or as much as tolerated by the patient.

On the first day of evaluation patients will first be interviewed to check GD diagnosis and screen other medical conditions that may exclude patients from the trial. The selected individuals will be randomly assigned to either naltrexone or placebo group; After that they will answer several questionnaires and have the first eye tracking assessment. Each individual will receive either placebo or naltrexone and be assessed 1 hour after drug administration.

After the first week patients will have the third eye tracking assessment, as well as several questionnaires On the next weeks patients will be constantly monitored for side effects and gambling symptoms.

On the twelfth week patients will have the fourth and last eye tracking assessment During the 12-week trial both groups will have psychoeducational sessions, on weeks 2,4,6 and 8. During sessions patients have access to audio-visual material and receive Self-help material, this intervention is based on Hodgins proposal (Hodgins DC et al, 2005).

Adherence will be verified by counting pills consumed by the patient. In the weeks without face-to-face medical assessment, patients will be evaluated by telephone interview to monitor adverse effects of medication. If the evaluator identifies a worrying adverse reaction, the patient will be advised to anticipate the face-to-face interview.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are:

  1. Men and woman aged 21 to 60 years;
  2. Female patients should be:

     * postmenopausal for at least one year, or;
     * are surgically unable to become pregnant (undergoing bilateral hysterectomy or oophorectomy or tubal ligation or otherwise unable to become pregnant), or;
     * be practicing an acceptable method of birth control (defined as hormonal contraceptives, spermicide plus barrier, a single vasectomized partner and / or intrauterine device);
  3. Have read and signed the informed consent form.

Exclusion Criteria:

* 1. Hypersensitivity to naltrexone or contraindication of naltrexone use; 2. Exposure to another pharmacological drug in the last 30 days; 3. Pregnancy or lactation; 4. Kidney dysfunction: Creatine serum > 133 mmol/L in men > 124 mmol/L in women, which correspond > 1,51 mg/dL e > 1,41 mg/Dl; 5. Liver dysfunction (aspartate transaminase (AST) and alanine transaminase (ALT) > 2times the upper limit of normal; 6. Cardiovascular disease, hypertension; 7. Lifetime history of bipolar disorder, Obsessive compulsive disorder, schizophrenia or any psychotic disorder, or depression (BDI> 30 points), clinically significant suicidality; 8. Lifetime history of drug (except nicotine) or alcohol; 9. Hematologic or immunologic dysfunction; 10. Subjects receiving psychoactive drugs, except sporadic use of benzodiazepines; 11. Simultaneous participation in other GD-related; 12. Lack of reliable contact information; 13. Illiteracy of other condition that difficult reading and understanding the study questionnaires and orientations; 14. Not having a cellphone line;

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Gambling Follow up scale (GFS) | Day 0 and day 84

SECONDARY OUTCOMES:
Gambling Self-Assessment Scale (G-SAS) | Day 0 and day 84
Gamblers´ Beliefs Questionnaires (GBQ) | Day 0 and day 84
Timeline Follow-Back Method, (TFB) | Day 0 and day 84
Barratt Impulsiveness Scale, version 11 | Day 0 and day 84
Social Adjustment Scale self-report version | Day 0 and day 84
Clinical Global Impression (CGI) | Day 0 and day 84

OTHER OUTCOMES:
Locus of control scale internal- external | Day 0,day 7, and day 84
Eye Tracking | Day 0, day 7 and day 84

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Altamirano LJ, Fields HL, D'Esposito M, Boettiger CA. Interaction between family history of alcoholism and Locus of Control in the opioid regulation of impulsive responding under the influence of alcohol. Alcohol Clin Exp Res. 2011 Nov;35(11):1905-14. doi: 10.1111/j.1530-0277.2011.01535.x. Epub 2011 May 13. PMID 21569055
- [Background] Anton RF, Moak DH, Waid LR, Latham PK, Malcolm RJ, Dias JK. Naltrexone and cognitive behavioral therapy for the treatment of outpatient alcoholics: results of a placebo-controlled trial. Am J Psychiatry. 1999 Nov;156(11):1758-64. doi: 10.1176/ajp.156.11.1758. PMID 10553740
- [Background] Brevers D, Cleeremans A, Bechara A, Laloyaux C, Kornreich C, Verbanck P, Noel X. Time course of attentional bias for gambling information in problem gambling. Psychol Addict Behav. 2011 Dec;25(4):675-82. doi: 10.1037/a0024201. Epub 2011 Jun 20. PMID 21688874
- [Background] Field M, Mogg K, Bradley BP. Cognitive bias and drug craving in recreational cannabis users. Drug Alcohol Depend. 2004 Apr 9;74(1):105-11. doi: 10.1016/j.drugalcdep.2003.12.005. PMID 15072814
- [Background] Field M, Mogg K, Zetteler J, Bradley BP. Attentional biases for alcohol cues in heavy and light social drinkers: the roles of initial orienting and maintained attention. Psychopharmacology (Berl). 2004 Oct;176(1):88-93. doi: 10.1007/s00213-004-1855-1. Epub 2004 Apr 8. PMID 15071718
- [Background] Galetti AM, Tavares H. Development and validation of the Gambling Follow-up Scale, Self-Report version: an outcome measure in the treatment of pathological gambling. Braz J Psychiatry. 2017 Jan-Mar;39(1):36-44. doi: 10.1590/1516-4446-2016-1911. Epub 2016 Nov 7. PMID 27828667
- [Background] Garbutt JC, Greenblatt AM, West SL, Morgan LC, Kampov-Polevoy A, Jordan HS, Bobashev GV. Clinical and biological moderators of response to naltrexone in alcohol dependence: a systematic review of the evidence. Addiction. 2014 Aug;109(8):1274-84. doi: 10.1111/add.12557. Epub 2014 May 23. PMID 24661324
- [Background] Grant LD, Bowling AC. Gambling Attitudes and Beliefs Predict Attentional Bias in Non-problem Gamblers. J Gambl Stud. 2015 Dec;31(4):1487-503. doi: 10.1007/s10899-014-9468-z. PMID 24871298
- [Background] Grant JE, Kim SW, Hartman BK. A double-blind, placebo-controlled study of the opiate antagonist naltrexone in the treatment of pathological gambling urges. J Clin Psychiatry. 2008 May;69(5):783-9. doi: 10.4088/jcp.v69n0511. PMID 18384246
- [Background] Hendershot CS, Wardell JD, Samokhvalov AV, Rehm J. Effects of naltrexone on alcohol self-administration and craving: meta-analysis of human laboratory studies. Addict Biol. 2017 Nov;22(6):1515-1527. doi: 10.1111/adb.12425. Epub 2016 Jul 14. PMID 27411969
- [Background] Hodgins DC. Implications of a brief intervention trial for problem gambling for future outcome research. J Gambl Stud. 2005 Spring;21(1):13-9. doi: 10.1007/s10899-004-1917-7. PMID 15789185
- [Background] Kim SW, Grant JE. An open naltrexone treatment study in pathological gambling disorder. Int Clin Psychopharmacol. 2001 Sep;16(5):285-9. doi: 10.1097/00004850-200109000-00006. PMID 11552772
- [Background] Kim SW, Grant JE, Adson DE, Shin YC. Double-blind naltrexone and placebo comparison study in the treatment of pathological gambling. Biol Psychiatry. 2001 Jun 1;49(11):914-21. doi: 10.1016/s0006-3223(01)01079-4. PMID 11377409
- [Background] Lahti T, Halme JT, Pankakoski M, Sinclair D, Alho H. Treatment of pathological gambling with naltrexone pharmacotherapy and brief intervention: a pilot study. Psychopharmacol Bull. 2010;43(3):35-44. PMID 21150845
- [Background] Lole L, Li E, Russell AM, Greer N, Thorne H, Hing N. Are sports bettors looking at responsible gambling messages? An eye-tracking study on wagering advertisements. J Behav Addict. 2019 Sep 1;8(3):499-507. doi: 10.1556/2006.8.2019.37. Epub 2019 Aug 26. PMID 31446764
- [Background] McGrath DS, Meitner A, Sears CR. The specificity of attentional biases by type of gambling: An eye-tracking study. PLoS One. 2018 Jan 31;13(1):e0190614. doi: 10.1371/journal.pone.0190614. eCollection 2018. PMID 29385164
- [Background] Mitchell JM, Tavares VC, Fields HL, D'Esposito M, Boettiger CA. Endogenous opioid blockade and impulsive responding in alcoholics and healthy controls. Neuropsychopharmacology. 2007 Feb;32(2):439-49. doi: 10.1038/sj.npp.1301226. Epub 2006 Oct 18. PMID 17047667
- [Background] Nestler EJ. From neurobiology to treatment: progress against addiction. Nat Neurosci. 2002 Nov;5 Suppl:1076-9. doi: 10.1038/nn945. PMID 12403990
- [Background] O'Brien CP, Volpicelli LA, Volpicelli JR. Naltrexone in the treatment of alcoholism: a clinical review. Alcohol. 1996 Jan-Feb;13(1):35-9. doi: 10.1016/0741-8329(95)02038-1. PMID 8837932
- [Background] Robinson TE, Berridge KC. Addiction. Annu Rev Psychol. 2003;54:25-53. doi: 10.1146/annurev.psych.54.101601.145237. Epub 2002 Jun 10. PMID 12185211
- [Background] Robinson TE, Berridge KC. Incentive-sensitization and addiction. Addiction. 2001 Jan;96(1):103-14. doi: 10.1046/j.1360-0443.2001.9611038.x. PMID 11177523
- [Background] Ruddock HK, Field M, Jones A, Hardman CA. State and trait influences on attentional bias to food-cues: The role of hunger, expectancy, and self-perceived food addiction. Appetite. 2018 Dec 1;131:139-147. doi: 10.1016/j.appet.2018.08.038. Epub 2018 Aug 29. PMID 30171914
- [Background] Sinclair JD. Evidence about the use of naltrexone and for different ways of using it in the treatment of alcoholism. Alcohol Alcohol. 2001 Jan-Feb;36(1):2-10. doi: 10.1093/alcalc/36.1.2. PMID 11139409
- [Background] Schultz W, Dayan P, Montague PR. A neural substrate of prediction and reward. Science. 1997 Mar 14;275(5306):1593-9. doi: 10.1126/science.275.5306.1593. PMID 9054347
- [Background] Vitaro F, Hartl AC, Brendgen M, Laursen B, Dionne G, Boivin M. Genetic and environmental influences on gambling and substance use in early adolescence. Behav Genet. 2014 Jul;44(4):347-55. doi: 10.1007/s10519-014-9658-6. Epub 2014 May 14. PMID 24824822
- [Background] Volpicelli JR, Alterman AI, Hayashida M, O'Brien CP. Naltrexone in the treatment of alcohol dependence. Arch Gen Psychiatry. 1992 Nov;49(11):876-80. doi: 10.1001/archpsyc.1992.01820110040006. PMID 1345133
- [Background] Wickelgren I. Getting the brain's attention. Science. 1997 Oct 3;278(5335):35-7. doi: 10.1126/science.278.5335.35. No abstract available. PMID 9340756
- [Background] Wilcockson TDW, Pothos EM. Measuring inhibitory processes for alcohol-related attentional biases: introducing a novel attentional bias measure. Addict Behav. 2015 May;44:88-93. doi: 10.1016/j.addbeh.2014.12.015. Epub 2014 Dec 27. PMID 25583563
- [Background] Yau YH, Potenza MN. Gambling disorder and other behavioral addictions: recognition and treatment. Harv Rev Psychiatry. 2015 Mar-Apr;23(2):134-46. doi: 10.1097/HRP.0000000000000051. PMID 25747926
- [Derived] Dowling N, Merkouris S, Lubman D, Thomas S, Bowden-Jones H, Cowlishaw S. Pharmacological interventions for the treatment of disordered and problem gambling. Cochrane Database Syst Rev. 2022 Sep 22;9(9):CD008936. doi: 10.1002/14651858.CD008936.pub2. PMID 36130734